CLINICAL TRIAL: NCT05809596
Title: HEAL-LAA: Post-Market Real World Outcomes in WATCHMAN FLX™ Pro Left Atrial Appendage Closure (LAAC) Device
Brief Title: HEAL-LAA Clinical Trial
Acronym: HEAL-LAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s2504
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation; Bleeding; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device Group (Other): WATCHMAN FLX Pro LAAC Device Implantation
  Interventions: Device: WATCHMAN FLX Pro LAAC Device

INTERVENTIONS:
Device: WATCHMAN FLX Pro LAAC Device — Treatment with a WATCHMAN FLX Pro Left Atrial Appendage Closure Device
  Other Names: Left Atrial Appendage Closure

SUMMARY:
The primary objective of this study is to collect real-world data on WATCHMAN FLX™ Pro Left Atrial Appendage Closure (LAAC) Device in patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of legal age to participate in the study.
* Subject has documented non-valvular atrial fibrillation (i.e., atrial fibrillation in the absence of moderate or greater mitral stenosis or a mechanical heart valve).
* Subject is clinically indicated for and is treated or attempted to be treated with a WATCHMAN FLX™ Pro device.
* Subject or legal representative is able to understand and willing to provide written informed consent to participate in the study.
* Subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

* Subject has a documented life expectancy of less than 6 months.
* Subject is currently enrolled in another investigational study, except if the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatment.
* Intracardiac thrombus is present.
* An atrial septal defect repair or closure device or a patent foramen ovale repair or closure device is present.
* The LAA anatomy will not accommodate a Closure Device.
* The patient has known hypersensitivity to any portion of the device material or the individual components such that the use of the WATCHMAN FLX™ Pro Device is contraindicated.
* Any of the customary contraindications for other percutaneous catheterization procedure (e.g., patient size too small to accommodate transesophageal echocardiography (TEE) probe or required catheters) or conditions (e.g., active infection, bleeding disorder) are present.
* There are contraindications to the use of anticoagulation therapy, aspirin, or P2Y12 inhibitor.
* Subject is of childbearing potential and is, or plans to become, pregnant during the time of the study (method of assessment per study physician's discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Kanj, MD, Principal Investigator — The Cleveland Clinic; Oluseun Alli, MD, Principal Investigator — Novant Health Heart & Vascular Institute
Locations (45):
- United States (45):
  - University of Alabama Medical Center, Birmingham, Alabama
  - Grandview Medical Center/ Affinity Cardiovascular Specialists, Birmingham, Alabama
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Scripps Memorial Hospital, La Jolla, California
  - Good Samaritan Hospital, Los Angeles, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - UC Health Memorial Hospital Central, Colorado Springs, Colorado
  - Cardiology Associates of Fairfield County, P.C., Norwalk, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Medical Center, Honolulu, Hawaii
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Heart and Vascular Hospital, Indianapolis, Indiana
  - University of Kansas Health System, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Health System, Kansas City, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Virtua Health, Marlton, New Jersey
  - Kaleida Health - Gates Vascular Institute, Buffalo, New York
  - Rochester General Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health Heart & Vascular Institute, Charlotte, North Carolina
  - Sanger Heart and Vascular Institute-Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Pinnacle Health at Harrisburg Hospital, Mechanicsburg, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Erlanger Health, Inc.,, Chattanooga, Tennessee
  - Baptist Memorial Hospital-Memphis / Stern Cardiovascular Foundation, Germantown, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Christus Trinity Mother Frances, Tyler, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy ( https://www.bostonscientific.com/en-US/data-sharing-requests.html).
Supporting Information: Study Protocol, SAP
Time Frame: 12 to 18 months following the end of the clinical trial. Estimated start Q4 2025, estimated end date Q4 2026-Q2 2027
Access Criteria: The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy ( https://www.bostonscientific.com/en-US/data-sharing-requests.html).
URL: https://www.bostonscientific.com/en-US/data-sharing-requests.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Analysis Subset: Initial 500 enrolled subjects
Period: Overall Study
Arm/Group | Primary Analysis Subset
Started | 500
45-Day Follow-up | 494
6-Month Follow-up | 474
Completed | 474
Not Completed | 26
Not completed — Death | 16
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Missed Visit | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Primary Analysis Subset
Number analyzed (Participants) | 500
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 188
  ≥ 75 years | 312
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 306
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 471
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race calculated for Non-Hispanic or Latino Ethnicity
  Participants
    number analyzed (Participants) | 471
    American Indian or Alaska Native | 1
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 2
    Black or African American | 20
    White | 441
    More than one race | 0
    Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 500

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint: The Rate of Device Leak >5 mm at 45-day Post-Implant TEE for the Primary Analysis Subjects
Description: Incomplete seal with peri-device gap > 5mm in the primary analysis subset implanted patients with 45-day TEE imaging (as assessed by the core lab).
Time Frame: 45 days
Population: Implanted primary analysis subjects with 45-day TEE imaging.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Analysis Subset: Initial 500 enrolled subjects (subjects who signed an approved Informed Consent Form, meet all clinical inclusion and no clinical exclusion criteria, and the WATCHMAN FLX Pro LAAC Device has been used for treatment and/or attempted to be used for treatment).
Arm/Group | Primary Analysis Subset
Number analyzed (Participants) | 404
Participants | 0

2. Primary Outcome: Primary Safety Endpoint: Composite Rate of All-cause Mortality, All Stroke, Systemic Embolism, and Major Bleeding for the Primary Analysis Subjects
Description: Composite CEC-adjudicated all-cause mortality, all stroke, systemic embolism, and major bleeding in the Intention to Treat (ITT) population at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Analysis Subset
Number analyzed (Participants) | 494
Participants | 54

ADVERSE EVENTS:
Time Frame: Study events are reported from enrollment through Day 180, with the exception of All-Cause Mortality which includes mortalities reported from enrollment through 6-month follow-up visit completion, or end of the 6-month visit window (210 days) when the visit was missed.
Arm/Group | Primary Analysis Subset
All-Cause Mortality (participants affected / at risk) | 16/500
Serious Adverse Events (participants affected / at risk) | 141/500
Other Adverse Events (participants affected / at risk) | 70/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Analysis Subset (N=500)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 13 (13)
Atrial flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 11 (13)
Cardiac failure congestive (Cardiac disorders) | 9 (10)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (13)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Catheter site discharge (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Device related thrombosis (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4)
Cystitis (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Pneumonia viral (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Pharyngeal perforation (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pericardial lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5)
Encephalopathy (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device extrusion (Product Issues) | 1 (1)
Device leakage (Product Issues) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Scalp haematoma (Vascular disorders) | 2 (2)
Subgaleal haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Analysis Subset (N=500)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Catheter site bruise (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 3 (3)
Catheter site pain (General disorders) | 2 (2)
Device related thrombosis (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Occult blood positive (Investigations) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 5 (5)
Haemorrhage (Vascular disorders) | 1 (1)
Scalp haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT05809596/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT05809596/SAP_002.pdf